CLINICAL TRIAL: NCT06615687
Title: Inverted T-shape Free Gingival Graft Versus Free Gingival Graft for Treatment of RT2/RT3 Gingival Recession Defects : a Randomized Clinical Trial
Brief Title: Inverted T-shape Free Gingival Graft for Treatment of RT2 / RT3 Gingival Recession Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Galal Fouad Mohamed Hafeez, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dgalal33724
Record Dates: First submitted 2024-09-14; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Gingival Recession
Keywords: Inverted T-shape Free Gingival Graft; Gingival Recession; Free Gingival Graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inverted T -Shape Free Gingival Graft (Experimental)
  Interventions: Procedure: Inverted T shape Free Gingival Graft
- Free Gingival Graft (Active Comparator)
  Interventions: Procedure: Free Gingival Graft

INTERVENTIONS:
Procedure: Inverted T shape Free Gingival Graft — the preparation of the recipient site commenced by making a horizontal incision at the mucogingival junction (MGJ) as well as two vertical incisions extending to the adjacent teeth and about 3-4 mm beyond the MGJ. A sharp split-thickness flap will be reflected, and the surfaces between these incisions will be de-epithelialized. Also, all the surfaces of the interdental papilla up to the lingual side will be de-epithelized using a 15c blade and microsurgical scissor .(Harvesting of the palatal donor site will be designed 2 mm away from the gingival margin using a template in the form of an inverted T-shape, taking into consideration the position of the greater palatine blood vessels at 5 mm. 2 mm is required for the width of the interproximal extension with 3 mm length to obtain an even thickness of 1-1.5 mm .
  Placement of the graft : The Inverted T FGG will be inserted between the teeth to cover interproximal tissue defect and sutured lingually into the lingual marginal gingiva
  Arms: Inverted T -Shape Free Gingival Graft
Procedure: Free Gingival Graft — Preparation of the recipient site :Following an intrasulcular incision, 2 mm-long horizontal incisions at the level of the CEJ will be performed bilaterally. From these, vertical releasing incisions will be placed in a diverging manner, extending well into the alveolar mucosa, a thin partial thickness flap will be subsequently raised then excised. The dimension of the resulting site will be measured to obtain a rectangular foil template .
  Harvesting of the Graft :Using the foil template, graft dimensions will be outlined in the palate adjacent to the premolars and first molar. A partial thickness graft consisting of epithelium and a thin layer of underlying connective tissue will be harvested (intended total thickness of graft: 1.5 mm), maintaining a distance of ≥2 mm to the maxillary teeth.
  Arms: Free Gingival Graft

SUMMARY:
The aim of this study is to compare the use of T-inverted shape Free Gingival Graft with Free Gingival Graft for improving the clinical attachment, gain partial root coverage, and improve Keratinized tissue width in recession type 2 /recession type 3 gingival recession defects .

Research question : In patients with RT2 / RT3 mandibular defects will the use of inverted T-shape free gingival graft differ from free gingival graft in Recession depth?

ELIGIBILITY:
Inclusion Criteria:

* Patients with RT2/RT3 gingival recession.
* Indication for FGG treatment at mandibular incisor area (i.e., difficulty or discomfort during oral hygiene; gingival margin mobility; high muscle attachment and/or frenum pull; shallow vestibule and gingival recession.
* KT width (KTW) < 2 mm.
* Ages 18-40 years old.
* Patients with healthy systemic condition (Brightman. 1994).
* Gingival and plaque index <10.
* Good oral hygiene (Wiesner et al. 2010).
* Accepts 6 months follow-up period (cooperative patients)

Exclusion Criteria:

* Smokers.
* Poor oral hygiene.
* Patient with a physical disability that hinders the upkeep of good oral hygiene measures.
* Intake of any medications known to affect gingival homeostasis or to interfere with wound healing.
* Pregnant or lactating women.
* RT1 gingival recession.
* Caries or non-carious cervical lesions at recipient sites.
* Severely malpositioned teeth.
* Teeth with residual probing depth ≥ 4 mm.
* Mobility ≥ 1 mm.
* Pervious periodontal surgery within the last 6 months before the start of the trial.
* Patients with active periodontal disease. -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Recession depth. | baseline, 1 month , 3 months and 6 months
  Will be measured as the distance from the CEJ to the most apical extension of the gingival margin.

SECONDARY OUTCOMES:
Width of keratinized gingiva . | baseline, 1 month , 3 months and 6 months
  Will be measured from the MGJ to the free gingival margin. The MGJ will be identified using the roll technique.
Recession width | baseline, 1 month , 3 months and 6 months
  Will be measured as the distance from mesial and distal papillae along the CEJ
Gingival thickness | baseline, 1 month , 3 months and 6 months
  An endodontic file and a 3 mm diameter silicon disc stop will be used to measure gingival thickness 2mm apical to the gingival border. The file will be inserted into the soft tissue with mild pressure, perpendicular to the mucosal surface, until a firm surface is felt. The silicon disc stop will be then pressed against the soft tissue, with the coronal border covering the soft tissue boundary.GT will be measured 2 mm apical from the gingival margin
Root coverage esthetic score | baseline, 1 month , 3 months and 6 months
  The RES system evaluated five variables 6 months following surgery: GM, marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment, and gingival color (GC). The clinical esthetic evaluation performed without magnification. Zero, 3, or 6 points were used for the evaluation of the position of the gingival margin, whereas a score of 0 or 1 point was used for each of the other variables.
The Distance between the contact point and the top of the papilla (DCP). | baseline, 1 month , 3 months and 6 months
  Measured as the distance between contact point and the tip of the papilla (DCP) in mms using UNC periodontal probe .
Probing Depth | baseline, 1 month , 3 months and 6 months
  The assessment of probing depth will be measured from the gingival margin to the bottom of the sulcus using a periodontal probe, rounded to the nearest millimeter.
Gingival Index | baseline, 1 month , 3 months and 6 months
  0 Normal gingiva.
  1. Mild inflammation.
  2. Moderate inflammation.
  3. Severe inflammation.
Plaque Index | baseline, 1 month , 3 months and 6 months
  0 No plaque in the gingival area.
  * 1 A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  * 2 Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  * 3 Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Galal Hafeez, Bachelor, Principal Investigator — Cairo University; Manar El-Zanaty, lecturer, Study Chair — Cairo University; Noha Ghallab, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Egypt